CLINICAL TRIAL: NCT01232192
Title: Study of Antenatal Model to Prevent Preterm Delivery: Early Detection and Treatment of Bacterial Vaginosis
Brief Title: Study of Antenatal Model to Prevent Preterm Delivery
Acronym: AACP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Showa University (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Fetal Maternal Divsion, Dept Obstetrics Gynecology, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AACP09
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2009-03

CONDITIONS: Preterm Delivery; Pregnant Women; Antenatal Care Model
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antenatal model (No Intervention)
  Interventions: Behavioral: antenatal model
- Antenatal Model (Experimental)
  Interventions: Behavioral: antenatal model

INTERVENTIONS:
Behavioral: antenatal model — Antenatal model is consisted of integrated efforts to lower preterm delivery rate through early detection and bacterial vaginal infection treatment:
  * Midwife training
  * Pregnant women campaigning
  * Early detection with self pH detection
  * Treatment of bacterial vaginosis
  Other Names: antenatal care model

SUMMARY:
The purpose of this study is to determine whether antenatal model in vaginosis are effective in preventing vaginal infection and preterm delivery

DETAILED DESCRIPTION:
The standard antenatal care nowadays can not answer for preterm delivery problems. Thus, comprehensive and proactive approach is needed for preventing preterm delivery. This antenatal model is consisted of midwife training, early detection of bacterial vaginosis, pregnant women campaign and self administered pH check

ELIGIBILITY:
Inclusion Criteria:

* 14- 18 week gestation pregnant women with or without any vaginal discharge
* singleton pregnancy, without any fetal or uterine anomaly

Exclusion Criteria:

* Any complication in pregnancy
* Any history of disease in pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
all preterm delivery | 37 weeks

SECONDARY OUTCOMES:
knowledge of midwife about preterm | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sungkar, MD, PhD, Principal Investigator — Dept Obstetrics Gynecology, Indonesia University
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Sungkar A, Purwosunu Y, Aziz MF, Pratomo H, Sutrisna B, Sekizawa A. Influence of early self-diagnosis and treatment of bacterial vaginosis on preterm birth rate. Int J Gynaecol Obstet. 2012 Jun;117(3):264-7. doi: 10.1016/j.ijgo.2012.01.007. Epub 2012 Mar 23. PMID 22445423